CLINICAL TRIAL: NCT00119184
Title: A Prospective Randomized Study to Examine the Success Rate of External Cephalic Version for Breech Presentation at Term Presentation: Spinal Analgesia Versus No Analgesia
Brief Title: Spinal Analgesia Versus No Analgesia: Study for External Cephalic Version
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Multiparas study terminated due to poor recruitment. Randomization revealed only after decision recorded on clinicaltrials.gov
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr Carolyn Weiniger, Hadassah HMO
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20-25/01/02-HMO-CTIL
Record Dates: First submitted 2005-07-03; First posted 2005-07-13 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2008-05

CONDITIONS: Breech Presentation
Keywords: anesthesia; breech; external cephalic version; spinal; success; anesthesia,spinal
MeSH Terms: conditions — Breech Presentation | interventions — Version, Fetal; Anesthesia, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- External cephalic version with spinal anesthesia (Experimental): External cephalic version with spinal anesthesia
  Interventions: Procedure: External cephalic version; Drug: spinal anesthesia
- External cephalic version without spinal anesthesia (Active Comparator): External cephalic version without spinal anesthesia
  Interventions: Procedure: External cephalic version

INTERVENTIONS:
Procedure: External cephalic version — 7.5 mg bupivacaine intrathecally
Drug: spinal anesthesia — spinal anesthesia
  Arms: External cephalic version with spinal anesthesia

SUMMARY:
The purpose of this study is to examine whether spinal anesthesia affects the chances of successful external cephalic version (ECV) of a breech presenting fetus.

Two study groups will be included; one will receive spinal anesthesia, the other will not. The non-spinal group will be permitted to cross over if ECV procedure is painful.

The main outcome is success of ECV.

DETAILED DESCRIPTION:
The rate of breech presentations in the general population of parturients has remained unchanged at 3%. However, the recent finding that the fetus has an increased morbidity during a vaginal delivery when compared with Cesarean section [1] has driven obstetricians towards the decision that all breech presentations will be delivered surgically. The morbidity of the mother with a breech presentation is not increased with a vaginal delivery; in fact the maternal morbidity associated with surgery is higher than after a vaginal delivery [2,3]. Subsequent pregnancies are automatically deemed high risk due to the presence of a uterine scar [4].

In an attempt to reduce the need for surgery with a breech presentation, the only option available in the current climate, where a vaginal delivery is out of the question, is to attempt to convert the fetal presentation from a breech to a vertex (head) presentation.

This technique may result in the premature onset of labor, which would require emergent surgery, and there is also a risk of placental abruption [5]. Following external cephalic version (ECV), the fetus may spontaneously return to the breech position. The success rates vary from 30% in nulliparous women, to 67% in multiparous women [6].

In an attempt to improve the success rates of ECV, authors have previously utilized regional anesthesia techniques [7-11]. Regional analgesia relaxes the stomach wall, and provides pain relief during the ECV procedure. The use of regional analgesia has claimed to increase the success rate of ECV to up to 80% [7]. However, other studies found no differences in success rates between the group which received regional analgesia and the group that did not [12]. All of these studies looked at women who have reached at least 36 weeks gestation. Despite the well-recognized differences in success rates between nulliparous and multiparous women, none of the studies that have examined regional analgesia with ECV have controlled for this factor in their studies. Thus the success rates, and any increase in success rates that is seen, may purely be a function of the number of multiparous women enrolled in the study.

This study will compare ECV separately in both a nulliparous and multiparous population, at term, and compare the success rates when spinal anesthesia is employed, versus no anesthesia. Success is defined as the conversion of a breech to vertex presentation.

Methods:

The study is prospective and randomized. Both nulliparous and multiparous women will be enrolled in the study, however each group will be randomized separately either to receive, or not receive, neuraxial (spinal) analgesia. Approximately 50 nulliparous and 50 multiparous women will be enrolled in each of the two groups. Randomization will be decided according to the final number of the patient's identity number (odd numbers will receive spinal analgesia, and even numbers will not receive analgesia). Written informed consent will be obtained prior to inclusion in the study.

All women will receive 20 mg nifedipine orally 30 minutes before the procedure according to hospital protocol. They will have continuous fetal heart rate monitoring.

After randomization, the spinal analgesia group (S) will receive 1000 cc Ringer's Lactate solution. Additional monitoring will include ECG, non-invasive blood pressure and pulse oximetry. In the sitting position, spinal anesthesia will be performed using a pencil-point needle. 7.5 mg plain bupivacaine (Astra) will be injected intrathecally. The patient will be reclined in a left lateral tilt, and the table will be adjusted in order to encourage the spreading of the anesthetic drug to the T6 level. Once anesthesia is attained, the ECV procedure will be performed.

The group assigned to receive no analgesia (N) will receive 1000 cc Ringer's Lactate solution prior to the ECV procedure. These women will be monitored in the same way as group S. ECV will be performed as usual. Women who are at an advanced stage of pregnancy, or have some other obstetric indication for delivery on the day of the ECV, will be offered their spinal analgesia with the addition of an epidural catheter (CSE-combined spinal epidural technique). This technique is part of regular daily anesthesia practise, and allows for the administration of additional analgesia after the effect of the spinal anesthesia has passed. This would be sufficient either for labor or for Cesarean section analgesia.

2 obstetricians, at least one of whom has experience with the procedure, will perform the ECV, with the aid of ultrasound surveillance. The ECV procedure will be halted if any of the following occurs: fetal bradycardia, placental abruption, and failure of ECV.

Women from group N who are unable to tolerate the procedure due to discomfort will be provided with regional analgesia, as described above.

Results:

The results will be analyzed on an intention to treat basis. Demographic data including age, parity, previous breech delivery, fetal size at 32 week ultrasound scan, and estimated amount of amniotic fluid will be collected and analyzed by ANOVA.

Data regarding success of ECV and complications will be analyzed using student t test and Chi square. Significance will be considered as p < 0.05.

Conclusion:

Success of the anesthesia-assisted ECV technique will be defined as a significant increase in the success rate of ECV, without a significant increase in the complication rate.

References:

1. Hannah ME, Hannah WJ, Hewson SA. Planned caesarean section versus planned vaginal birth for breech presentation at term: a randomized multicentre trial Term Breech Collaborative Group. Lancet 2000 Oct; 356 (9239): 1368-9.
2. Sanchez-Ramos L, Wells TL, Adair CD. Route of breech delivery and maternal and neonatal outcomes. Int J Gynecol Obstet 2001 Apr;73(1):7-14.
3. Jackson N, Paterson-Brown S. Physical Sequelae of caesarean section. Best Pract Res Clin Obstet Gynecol 2001 Feb; 15 (1):49-61.
4. Mozurkewitch EL, Hutton EK. Elective repeat cesarean section versus trial of labor: a metanalysis of the literature from 1989-1999. Am J Obstet Gynecol 2000 Nov;183 (5): 1187-97.
5. Kasule J, Chimbria TH, Brown IM. Controlled trial of external cephalic version. Br J Obstet Gynaecol 1985;92:14-8.
6. Ezra Y, Elram T, Plotkin V, Elchalal U. Significance of success rate of external cephalic versions and vaginal breech deliveries in counseling women with breech presentation at term. Eur J Obstet Gynecol Reprod Biol 2000 May;90 (1):63-6.
7. Birnbach DJ, Matut J, Stein DJ et al. The effect of intrathecal analgesia on the success of external cephalic version. Anesth Analg 2001 Aug; 93(2):410-3.
8. Mancuso K, Yancey MK, Murphy JA et al. Epidural analgesia for cephalic version: a randomized trial. Obstet Gynecol 2000 may;95(5):648-51.
9. Neiger R, Hennessy MD, Patel M. Reattempting failed external cephalic version under epidural anesthesia. Am J Obstet Gynecol 1998 Nov;179(5):1136-9.
10. Schorr SJ, Speights SE, Ross EL et al. A randomized trial of epidural anesthesia to improve external cephalic version success. Am J Obstet Gynecol 1997 Nov;177(5):1133-7.
11. Carlan SJ, Dent JM, Huckaby et al. The effect of epidural anesthesia on the safety and success of external cephalic version at term. Anesth Analg 1994 Sept;79(3):525-8.
12. Dugoff L, Stamm CA, Jones OW 3rd et al. The effect of spinal anesthesia on the success rate of external cephalic version: a randomized trial. Obstet Gynecol 1999 Mar;93(3):345-9.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* 37 + weeks gestation
* No previous attempt at ECV in this pregnancy
* No fetal abnormality

Exclusion Criteria:

* No previous uterine surgery
* Any contraindication for vaginal delivery
* Contra-indications to regional analgesia: uncorrected hypovolemia, coagulopathy (including anti-coagulants but not low-dose [100mg] aspirin), infection or inflammation of the skin overlying the lumbar area, raised intra-cranial pressure, hypersensitivity to amide local anesthetic agents.
* Patient refusal for regional analgesia
* Previous history of meningitis, neuropathy, or severe back pain with neurological radiation
* Poor communication (no Hebrew or English spoken, deafness, blindness, serious intellectual impairment or psychiatric disorder)
* Morbid obesity

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2002-10; Primary Completion 2006-03 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Conversion of a breech to a vertex presentation | 4-6 years

SECONDARY OUTCOMES:
Complications associated with ECV: Premature rupture of membranes, Contractions, Placental abruption, Fetal distress, Pain score during procedure (VAS Scale 0 = no pain, 10 = severe pain). | 4-6 years
Complications associated with analgesia: Severe maternal hypotension (>20 reduction in systolic BP), Fetal distress (prior to performance of ECV), Post Dural Puncture Headache, Failure of analgesia. | 4-6 years
Inability to perform procedure due to maternal distress or discomfort. | 4-6 years
Mode of delivery and date from the ECV. | 4-6 years

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn F Weiniger, MB ChB, Principal Investigator — Dept Anesthesiology, Hadassah Hebrew University Medical School
Locations (1):
- Hadassah Hebrew University Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Weiniger CF, Ginosar Y, Elchalal U, Sela HY, Weissman C, Ezra Y. Randomized controlled trial of external cephalic version in term multiparae with or without spinal analgesia. Br J Anaesth. 2010 May;104(5):613-8. doi: 10.1093/bja/aeq053. Epub 2010 Mar 25. PMID 20338954
- [Derived] Weiniger CF, Ginosar Y, Elchalal U, Sharon E, Nokrian M, Ezra Y. External cephalic version for breech presentation with or without spinal analgesia in nulliparous women at term: a randomized controlled trial. Obstet Gynecol. 2007 Dec;110(6):1343-50. doi: 10.1097/01.AOG.0000295605.38175.7b. PMID 18055730